CLINICAL TRIAL: NCT04582383
Title: A Randomized, Double-Blind, Multi-Center Comparative Effectiveness Study of Spironolactone Versus Doxycycline Hyclate for the Treatment of Acne in Women
Brief Title: Comparative Effectiveness Study of Spironolactone Versus Doxycycline for Acne
Acronym: SD-ACNE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R34AR074733-01A1 (NIH)
Record Dates: First submitted 2020-09-30; First posted 2020-10-09 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Acne
Keywords: spironolactone; doxycycline
MeSH Terms: conditions — Acne Vulgaris | interventions — Spironolactone; Doxycycline

STUDY DESIGN:
Intervention Model Description: 175 participants will be randomized to treatment with spironolactone 100mg/day and 175 participants will be randomized to treatment with doxycycline hyclate 100mg/day.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spironolactone (Experimental): In this arm, participants will receive spironolactone 100mg/day for the entirety of the study. To maximize the generalizability of the study, participants will be allowed to continue their current topical regimen as long as no changes were made in the 4 weeks prior to randomization. No additions to their topical regimen may be made during the study period.
  Interventions: Drug: Spironolactone
- Doxycycline hyclate (Active Comparator): This arm is an active-comparator arm in which participants will receive doxycycline hyclate 100mg/day for the entirety of the study. To maximize the generalizability of the study, participants will be allowed to continue their current topical regimen as long as no changes were made in the 4 weeks prior to randomization. No additions to their topical regimen may be made during the study period.
  Interventions: Drug: Doxycycline Hyclate

INTERVENTIONS:
Drug: Spironolactone — Dispensation of spironolactone according to the arm description.
  Arms: Spironolactone
Drug: Doxycycline Hyclate — Dispensation of doxycycline hyclate according to the arm description.
  Arms: Doxycycline hyclate

SUMMARY:
Acne is common illness of adolescents and young adults which is associated with substantial morbidity. While topical treatments are often sufficient for mild acne, moderate to severe acne often requires treatment with systemic medications such as oral antibiotics, hormonal therapies such spironolactone, and isotretinoin. Sebum overproduction is fundamental to the pathogenesis of acne with associated disordered keratinization and subsequent microbial colonization and inflammation resulting in the clinical manifestations of acne. Given the influence of hormones on sebum production, therapies that address these underlying hormonal factors such as spironolactone and oral contraceptive pills represent an underutilized treatment option for women with acne and could help decrease the use of long-term oral antibiotics in this patient population. The purpose of this trial is to evaluate the comparative effectiveness of spironolactone versus doxycycline hyclate (tetracycline class antibiotic) for women with acne.

ELIGIBILITY:
Inclusion Criteria:

* Female sex assigned at birth
* Age 16-40 years old
* Acne defined as at least 10 inflammatory papules or pustules and an Investigator's Global Assessment (IGA) score of at least 2 as measured by the Comprehensive Acne Severity Scale
* Not currently pregnant or planning to become pregnant

Exclusion Criteria:

* Pregnancy
* Heart disease
* Renal disease
* Liver disease
* Orthostatic hypotension
* Addison's disease
* History of hyperkalemia
* Allergy to tetracycline-class antibiotic
* Allergy to spironolactone
* Concomitant use of medications known to interact with spironolactone or doxycycline or that may increase the risk for hyperkalemia, including angiotensin-converting enzyme inhibitors, angiotensin receptor blockers, eplerenone, nonsteroidal anti-inflammatory drugs, and digoxin.
* Treatment with spironolactone, an oral antibiotic, laser, photodynamic therapy, or chemical peel within the past 4 weeks
* Treatment with isotretinoin within the past 3 months
* Sebacia laser treatment within the past 12 months

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2026-02-17 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Absolute change in inflammatory lesion count | Baseline to Week 16
  Difference in change in inflammatory lesion count between those randomized to spironolactone versus doxycycline hyclate

SECONDARY OUTCOMES:
Percentage achieving Investigator Global Assessment (IGA) Success (IGA grade of clear or almost clear; grade 0 or 1) | Baseline to Week 8, and Week 16
  Difference in percentage achieving IGA success between those randomized to spironolactone versus doxycycline hyclate
Change in comedonal lesions | Baseline to Week 8, and Week 16
  Difference in change in comedonal lesions between those randomized to spironolactone versus doxycycline hyclate
Change in Acne-QoL, an acne-specific quality of life measure | Baseline to Week4, Week 8, Week 12, and Week 16
  Difference in change in Acne-QoL score between those randomized to spironolactone versus doxycycline hyclate. There are 4 subscales: self perception, scored 0-30; role social, scored 0-24; role-emotional, scored 0-30; and acne symptoms, scored 0-30. Higher scores indicate better quality of life.
Change in Dermatology Life Quality Index (DLQI), a dermatology-specific quality of life measure | Baseline to Week4, Week 8, Week 12, and Week 16
  Difference in change in DLQI score between those randomized to spironolactone versus doxycycline hyclate. Scores range from 0-30, with lower scores indicated better quality of life.
Patient global assessment | Baseline to Week4, Week 8, Week 12, and Week 16
  Difference in change in patient global assessment scores between those randomized to spironolactone versus doxycycline hyclate.
Percentage on any topical medication at baseline who discontinued at least one of these topical medications (i.e. topical retinoid, benzoyl peroxide, and topical antibiotic) | Baseline to Week 16
  Difference between those randomized to spironolactone versus doxycycline hyclate

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Johnson Dermatology, Fort Smith, Arkansas
  - University of California San Francisco, San Francisco, California
  - Cura Clinical Research, Sherman Oaks, California
  - University of Miami, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - New York University, New York, New York
  - Northwell Health, North New Hyde Park, New York
  - Dermatologists of Central States, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Cyn3rgy Research, Gresham, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Arlington Research Center, Arlington, Texas
  - North Texas Center for Clinical Research, Frisco, Texas
  - CCS Texas, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available to research teams within 1 year following study completion.
Supporting Information: Study Protocol, SAP
Time Frame: 1 year following study completion